CLINICAL TRIAL: NCT05122481
Title: Vitamin C 4 Care Homes: a Pilot and Feasibility Study to Assess Daily Vitamin C Requirement of Care Home Residents
Brief Title: Vitamin C 4 Care Homes
Acronym: VITA-C4CARE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Aberdeen (Other)
Collaborators: University of Otago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2-061-21; 296819 (Other: IRAS)
Record Dates: First submitted 2021-09-15; First posted 2021-11-16 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Hypovitaminosis; Vitamin C Abnormal
Keywords: Vitamin C; Care home; Hypovitaminosis
MeSH Terms: conditions — Avitaminosis | interventions — Ascorbic Acid

STUDY DESIGN:
Intervention Model Description: This is a pilot dose-finding study comprising 20 older people ENRICH listed care home residents (aged 65+) with capacity.
Masking Description: Randomized number allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Care home residents (Experimental): On the test days, the participant will be asked to provide a urine sample before taking the supplement, this sample will be used as a baseline and assessed for Vitamin C and creatinine/protein and specific gravity, with the same testing strips as mentioned above. Once collected, the participant will be provided with a drink containing an increasing daily dose of vitamin C (0 - 500 mg). A second urine sample will then be collected approx. 3 - 4 hours later to assess the extent of vitamin C excretion in urine with an increase in vitamin C supplement. Another urine test strip will also be used to determine creatinine concentrations, the presence of albumin/protein, and specific gravity (to determine urine concentration). Up to 3 days will be allowed between daily testing to allow for long weekends, absences, illness, etc. Therefore, the participants are expected to complete the study within 4 weeks.
  Interventions: Dietary Supplement: Vitamin C

INTERVENTIONS:
Dietary Supplement: Vitamin C — Vitamin C (also known as ascorbic acid and ascorbate) is a vitamin found in various foods and sold as a dietary supplement.Vitamin C is a water-soluble vitamin, with dietary excesses not absorbed, and excesses in the blood rapidly excreted in the urine, so it exhibits remarkably low acute toxicity. More than one gram may cause indigestion, flatulence and stomach pain.
  Other Names: Ascorbic Acid; Vit. C; ascorbate

SUMMARY:
Older people in care homes are one of the most vulnerable groups with respect to risk, morbidity and mortality of severe coronavirus disease-2019 (COVID-19). In the UK, almost half (47%) of all COVID-19 deaths occurred in care homes. The World Health Organization (WHO) has highlighted vitamin C as an adjunctive therapy with biological plausibility for people with severe COVID-19. Previous research has indicated that up to 40% of care home residents in the UK are deficient in vitamin C, an essential immune supportive nutrient. This is a 10-fold higher deficiency level than that reported in community dwelling older people in the UK government's National Diet and Nutrition Survey.

Due to lack of robust pharmacokinetic data in older people, the intake required to optimise the vitamin C status of this cohort is not yet known and may be higher than that for healthy adults; some have estimated as high as 400 mg/d (the current UK recommended nutrient intake (RNI) or vitamin C is 40 mg/d, which is sufficient to prevent deficiency, but not enough for optimal/saturating vitamin C status). Thus, this pilot and feasibility study will assess the intake requirements of care home residents for optimal vitamin C status. The purpose is to provide essential data for a future clinical trial assessing the efficacy of optimal vitamin C supplementation for risk, severity, and duration of respiratory infections in this population who are at risk of such infections.

DETAILED DESCRIPTION:
This is a pilot dose-finding study comprising 20 older people ENRICH-listed care home residents (aged 65+). The feasibility of a larger study and a future trial recruitment will also be assessed.

The investigators will invite care homes to participate in the study by approaching care homes that have expressed interest in hosting research studies as research sites via care home network ENRICH (https://enrich.nihr.ac.uk/joining-the-network/). Flyers will also be provided (VitaC4Care_ V.3 _14.09.21_ Flyer) to raise interest.

Each participant, with the assistance of a care home staff member, will complete a two-part questionnaire at the beginning of the study and at the end. The first part of the questionnaire will include recordings of age, weight/height, date of admission to care home and date of completion of the present questionnaire, co-morbidities (specifically hypertension, diabetes, previous cerebrovascular accident or myocardial infarction, arthritis, Chronic obstructive pulmonary disease or asthma, active malignancy, and type), regular medication (specifically omeprazole, diabetic medication and type, aspirin, diuretics and type, and statins). The first-part questionnaire will include free text spaces for the addition of other comorbidities or medications not mentioned above. For the second part of the questionnaire, the participant will be required to complete a symptom record for the following symptoms: arthralgia (lay language as per patient questionnaire: sore joints), myalgia (sore muscles) ankle edema (puffy ankles), loss of appetite, peripheral paresthesia (pins and needles at hands or legs), dizziness, shortness of breath, malaise (tiredness), low mood, irritability. The participant will be required to state how often they experience these symptoms on a scale from 1 (Never) to 5 (All the time). The same questionnaire will be offered to the participants at the end of the study and symptom improvement, or deterioration will be recorded on a numerical scale. Furthermore, each participant (assisted by care home staff) will provide twelve urine samples over the course of up to four weeks which will be analysed for vitamin C content using a urine vitamin C test strip (VitaChek-C, Teco Diagnostics, USA) and creatinine/protein/Specific Gravity ((HomeHealth, UK). There will be six designated test days and the rest of the study period will be made up of break days when no samples will be collected. After each test day, three break days will be allowed to ensure participant comfort. If on a "testing" day, a second urine sample is not obtained, the same supplement concentration will be provided on the next "testing" day to ensure data completion.

On the test days, the participant will be asked to provide a urine sample before taking the supplement (Vitamin C 5000, NutriVital Food Supplement, made in UK by NutriVital Health, nutrivital.co.uk), this sample will be used as a baseline and assessed for Vitamin C and creatinine/protein and specific gravity, with the same testing strips as mentioned above. Once collected, the participant will be provided with a drink containing an increasing daily dose of vitamin C (0 - 500 mg; see study schedule in 3.2). The supplement will be encapsulated and either consumed as a pill or dissolved in a room temperature water drink prior to consumption.

A second urine sample will then be collected approx. 3 - 4 hours later to assess the extent of vitamin C excretion in urine with an increase in vitamin C supplement. Another urine test strip will also be used to determine creatinine concentrations (to standardize vitamin C values), presence of albumin/protein (to determine kidney function) and specific gravity (to determine urine concentration).

The absence of vitamin C in the urine or minimal change in excretion indicates that the blood is not yet saturated. In which case, the next dose will be given the following day.

Additional information on vitamin C dietary intake will be estimated by accessing the weekly care home menu, individual choice of menu and record of drink/food brought to care home residents by visitors. Information on demographics, length of time in care home, co-morbidities, and medications as documented in the care home records will also be collected.

This pilot study will provide the following information for power calculations for a larger study (future clinical trial):

1. the proportion of eligible older adults with inadequate vitamin C status
2. the minimum dose of vitamin C required to optimize plasma vitamin C status in this cohort To achieve the secondary objectives, information on the key aspects of feasibility for a larger study will be collected as described in the secondary objectives section (future clinical trial).

At the end of the study, a questionnaire will be disseminated to participants, their carers, relevant managers and care home staff to assess the willingness to participate in a bigger research trial and to identify any issues to be addressed to gain support for such an intervention trial. The questionnaire will be sent out to 31 individuals and will not collect any identifiable data. The recipient will have state their level of involvement to the study (e.g. participant, care home staff, care home manager, other (with free text).

ELIGIBILITY:
Inclusion Criteria:

1. Resident in a care home
2. Aged ≥65 years

Exclusion Criteria:

1. Unable to give fully informed consent, e.g. due to severe dementia
2. Any health conditions precluding collection of fresh urine samples (e.g. urinary catheter)
3. Active (acute) respiratory infection
4. Currently taking vitamin C containing supplements at greater than the recommended dietary intake (40 mg/d)

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-01-15 (Estimated); Primary Completion 2023-07-30 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants reporting hypovitaminosis symptoms by end of study | 6 days
  Any symptoms which participants report which are listed in vitamin C overdose signs and symptoms

SECONDARY OUTCOMES:
The feasibility of undertaking a study with this group of older people in a care home setting. | 2 months
  Successful recruitment and completion of study procedures to 100% target

CONTACTS AND LOCATIONS:
Locations (1):
- University of Aberdeen, Aberdeen, Aberdeen City, United Kingdom

IPD SHARING:
Plan to Share IPD: No